CLINICAL TRIAL: NCT02684825
Title: Detection of Silent Atrial Fibrillation aFter Ischemic StrOke (SAFFO) Guided by Implantable Loop Recorder. Multicentre Italian Trial Based on Stroke Unit Network With Paired Cardio-Arrhythmology Units (Italian Neurocardiology Unit Network)
Brief Title: Detection of Silent Atrial Fibrillation aFter Ischemic StrOke
Acronym: SAFFO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danilo Toni (Other)
Collaborators: Associazione Italiana Aritmologia e Cardiostimolazione (A.I.A.C.) - Stefano Strano, MD (Unknown); Boehringer Ingelheim (Industry); Medtronic Italia S.p.A. (Unknown); Bayer S.p.A (Unknown)
Responsible Party: Sponsor-Investigator, Danilo Toni, Director, Emergency Department Stroke Unit - Associate Professor of Neurology, Azienda Policlinico Umberto I
Organization: Azienda Policlinico Umberto I (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APUmbertoI
Record Dates: First submitted 2016-02-02; First posted 2016-02-18 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Ischemic Stroke; Cerebral Infarction; Brain Ischemia; Brain Infarction; Cerebrovascular Disorders; Brain Disease; Central Nervous System Diseases; Nervous System Diseases; Cardiac Arrhythmias
Keywords: Stroke; ischemic stroke; atrial fibrillation; continuous cardiac monitoring; insertable cardiac monitoring; implantable loop recorder; antithrombotics; anticoagulants; stroke subtype; atherothrombotic stroke; lacunar stroke
MeSH Terms: conditions — Ischemic Stroke; Cerebral Infarction; Brain Ischemia; Brain Infarction; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Arrhythmias, Cardiac; Stroke; Atrial Fibrillation; Stroke, Lacunar

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous plus standard cardiac monitoring (Experimental): Continuous cardiac monitoring by Reveal LINQTM- LNQ11 Internal Loop Recorder (ILR) plus standard cardiac monitoring
  Interventions: Device: Reveal LINQTM- LNQ11 Internal Loop Recorder plus standard cardiac monitoring
- Standard cardiac monitoring (No Intervention): Routine cardiac monitoring with follow-up at the same frequency, but with no Implantable Loop Recorder

INTERVENTIONS:
Device: Reveal LINQTM- LNQ11 Internal Loop Recorder plus standard cardiac monitoring — Reveal LINQTM- LNQ11 continuously monitors cardiac electric activity for up to three years.
  Other Names: Reveal LINQTM- LNQ11
  Arms: Continuous plus standard cardiac monitoring

SUMMARY:
The primary objective of this study is to evaluate whether, in patients with first-ever atherothrombotic or lacunar stroke without any previous history of atrial fibrillation (AF)/atrial flutter (AFL)/atrial tachycardia (AT), the detection of AF/AFL/AT (silent or symptomatic) by using a continuous cardiac rhythm monitoring with implantable loop recorder (ILR) during the first 12 months of observation is higher than the detection by using a standard cardiac monitoring (physical exam, 12-lead electrocardiogram [ECG] at baseline, 3, 6, and 12 months and Holter ECG at 3 months) in the same period of time.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is associated with a high risk of stroke and its prevalence increases in subjects aged ≥65 years. After an ischemic stroke, the use of standard monitoring methods may underestimate the detection rate of AF. Recent studies demonstrated a fourfold to sixfold increase in the detection of AF with prolonged ECG monitoring as compared to standard cardiac monitoring in patients with cryptogenic stroke. Hence, it is very likely that even patients having a first atherothrombotic or lacunar stroke with high burden of vascular risk factors are exposed to increased risk of developing AF in the subsequent years and AF may be the cause underlying possible recurrent strokes.

SAFFO trial has the objective to evaluate the detection of AF or atrial flutter (AFL) as first diagnosis by implantable loop recorder (ILR) in patients with first-ever atherothrombotic or lacunar stroke. Patients with recent (30-60 days after symptom onset) diagnosis of first-ever atherothrombotic or lacunar ischemic stroke who fulfill inclusion criteria will be randomized to either continuous cardiac monitoring using an ILR plus standard cardiac monitoring (intervention arm) or standard cardiac monitoring alone (control arm) with a ratio of 1:1. The hypothesis is that the detection of of AF/AFL by using ILR will be higher than that observed by using standard cardiac monitoring. Secondary and tertiary objectives of the study include exploratory analyses on the incidence of recurrent strokes and different stroke subtypes and on the reduction of stroke risk and death from all causes in all study patients, in the two randomization groups and, in particular, in patients treated with antiplatelet therapy versus those treated with oral anticoagulant (OAC) therapy, the latter being implemented and guided by the detection of clinically meaningful episodes of AF/AFL/AT using ILR compared with standard cardiac monitoring. Moreover, this study has the objective to evaluate a clinical, neuroimaging, and echocardiographic profile predictive of AF/AFL/AT first diagnosis and stroke recurrence.

SAFFO is a prospective, multicenter, randomized, controlled, open-label trial with blinded assessment of outcome measures. Diagnosis of atherothrombotic and lacunar etiology will be defined according to TOAST (trial of ORG 10172 in acute stroke treatment) / CCS (Causative Classification System for ischemic stroke) classification criteria and standard diagnostic protocols that have to be fulfilled before randomization (medical history; risk factors; symptoms; cerebral magnetic resonance [MR] and/or CT; 12-lead ECG and/or Holter ECG and/or other standard heart rhythm monitoring procedure; transthoracic and/or transoesophageal echocardiogram; intra- and extracranial vessel ultrasonography and/or CT-Angiography and/or MR- Angiography, also in order to rule out non-atherosclerotic vasculopathies; thrombophilic/hematologic screening if hypercoagulability states or other hematologic disorders are suspected).

ILR (Medtronic Reveal LINQTM- LNQ11REVEAL LinQ) implantation will be performed within 8 days after randomization and will allow a continuous monitoring by single-lead ECG registration for 3 years. Standard cardiac rhythm monitoring includes: detailed data collection on any possible patient's symptom suggestive of AF/AFL/AT, physical exam including cardiovascular examination, 12-lead ECG, and 24-hour Holter ECG performed at 3-month follow-up visit.

If positive, SAFFO trial could have important clinical implications in terms of changing the standard diagnostic protocol in patients with atherothrombotic and lacunar stroke, and of increasing the shift of secondary prevention treatment from antiplatelet to anticoagulant therapy when indicated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years old in the presence of at least one of the following vascular risk factors: hypertension; diabetes; vascular disease (previous myocardial infarction, peripheral arteriopathy).
* Age between 60 and 64 years old in the presence of at least two of the following vascular risk factors: hypertension; diabetes; vascular disease (previous myocardial infarction, peripheral arteriopathy); smoking.
* Recent (30-60 days after symptom onset) diagnosis of first-ever ischemic stroke. Ischemic stroke is defined as an event characterized by the sudden onset of acute focal neurological symptoms, MR or CT findings consistent with ischemic stroke, and no evidence of other neurological disorders clinically or radiographically to explain. Patients with reversible neurological deficit within 24 hours (clinical TIA), but with a cerebral injury of ischemic origin visible on neuroimages and corresponding to patient symptoms, have to be classified as having an ischemic stroke and considered for the study.
* Diagnosis of atherothrombotic and lacunar etiology, defined according to the TOAST classification criteria and standard diagnostic protocols that have to be fulfilled before randomization (medical history; risk factors; symptoms; cerebral MR and/or CT; 12-lead ECG and/or Holter ECG and/or other standard heart rhythm monitoring procedure; transthoracic and/or transoesophageal echocardiogram; intra- and extracranial vessel ultrasonography and/or CT-Angiography and/or MR-Angiography, also in order to rule out non-atherosclerotic vasculopathies; thrombophilic/hematologic screening if hypercoagulability states or other hematologic disorders are suspected).
* Neurological severity in terms of functional dependency defined as mRS (modified Rankin Scale) score ≤3.
* Written informed consent.

Exclusion Criteria:

* TIA without evidence of cerebral infarction on neuroimaging corresponding to patient symptoms.
* Diagnosis of cardioembolic stroke based on medical history and cerebral/cardiological/vascular diagnostic evaluation (e.g., evidence of a high-risk emboligenic source from the heart or aortic arch such as: left ventricle or atrium thrombus or "smoke", emboligenic valvular lesions, or emboligenic tumor, patent foramen ovale [PFO] associated with a possible venous thromboembolic source and hence eligible for oral anticoagulant [OAC] therapy, aortic arch plaques having >3 mm thickness or containing mobile components, or any other high-risk embolic lesion).
* Diagnosis of ischemic stroke of different etiopathogenesis, for example due to non-atherosclerotic vasculopathies, hypercoagulability states (diagnosed by a thrombophilic screening) or other hematologic disorders; or diagnosis of cryptogenic stroke.
* Previous documented history of atrial fibrillation (AF) or atrial flutter (AFL)
* History of untreated hyperthyroidism
* History of myocardial infarction <1 month before the study screening visit
* Valvular disease requiring immediate surgical intervention
* Recent (<6 months before the study screening visit) cardiac surgery
* Other conditions associated with an increased risk of AF: sick sinus syndrome, recent (<14 days before the study Screening visit) surgery; current infections
* Permanent indication for anticoagulation
* Contraindications to OAC therapy
* Stroke associated with severe functional disability defined as mRS>3
* Hear failure associated with severe ventricular dysfunction and ejection fraction ≤40%
* Indication for pacemaker or defibrillator implant
* Any condition that, in the opinion of the investigator, could make non feasible or hazardous patient's participation in the study or any condition that could compromise the completion of patient's participation in terms of follow-up visits (for example, diseases associated with a poor prognosis and life expectancy <1 year).
* Severe renal failure or liver disease
* Participation in any other clinical trial that can interfere with the objectives of the study
* Poor patient's compliance that could compromise his/her correct participation in the study
* Patient's refusal to give his/her informed consent for the participation in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 317 (Actual)
Dates: Start 2015-10; Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Detection rate of AF/AFL/AT within 12 months | 12 months
  Episodes of AF/AFL/AT will be adjudicated by an independent committee of cardiologists blinded to randomization arm

SECONDARY OUTCOMES:
Incidence of ischemic stroke recurrence and incidence of the different ischemic stroke subtypes | 36 months
  Stroke subtypes will be adjudicated by an independent committee of neurologists blinded to randomization arm
Reduction of the risk of ischemic stroke and death from all causes | 36 months
  Reduction of the risk of ischemic stroke and death from all causes will be evaluated in particular in patients treated with antiplatelet therapy versus those treated with OAC therapy, the latter being implemented and guided by the detection of clinically meaningful episodes of AF/AFL/AT using ILR compared with standard cardiac monitoring

OTHER OUTCOMES:
Rate of asymptomatic/symptomatic episodes of AF/AFL/AT | 36 months
Use of oral anticoagulant (OAC) drugs | 36 months
  Percentage of subjects who will use OAC drugs at the 36-month follow-up visit
Use of antiarrhythmic drugs | 36 months
  Percentage of subjects who will use antiarrhythmic drugs at the 36-month follow-up visit
Time from AF/AFL/AT detection to the change of secondary prevention treatment from antiplatelet to OAC therapy | 36 months
Burden of AF/AFL/AT and relative clinical, imaging, and treatment associations | 36 months
Progression of the cerebrovascular damage | 36 months
  Progression of cerebrovascular damage will be evaluated in terms of increase of silent infarct number, leukoaraiosis/white matter hyperintensity, microbleeds, dilated perivascular spaces, and brain atrophy measured on MR
Progression of possible cognitive impairment | 36 months
  Minimental State Examination (MMSE) and Montreal Cognitive Assessment (MoCA) are scales that will be used to measure cognitive functions
Health outcome as evaluated by ED-5D-3L Questionnaire | 36 months
  EQ-5D-3L (visual analog scale, VAS) quality of life score is a continuous measure of quality of life ranging from 0 (worst) to 100 (perfect health)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Policlinico Umberto I, Rome, Italy